CLINICAL TRIAL: NCT06998849
Title: The Impact of Intraoperative Change in the Body Temperature on the Perfusion Index: : A Cross-sectional Study
Brief Title: The Impact of Intraoperative Change in the Body Temperature on the Perfusion Index
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS143/2024
Record Dates: First submitted 2025-04-04; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-04

CONDITIONS: Perfusion Index; Hypothermia; Anesthesia
Keywords: Cross sectional; Observational; Hypothermia; Anaesthesia; Anesthesia; General Anaesthesia; General Anesthesia; General surgery
MeSH Terms: conditions — Hypothermia | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients undergoing general surgery: Adult patients undergoing elective general surgery
  Interventions: Diagnostic Test: Perfusion index

INTERVENTIONS:
Diagnostic Test: Perfusion index — The perfusion index (PI) is defined as the ratio of pulsatile light absorption to continuous light absorption, denoted as AC/DC. Initially used as a quality signal indicator in pulse oximetry, PI has increasingly been recognized for its potential in non-invasive hemodynamic monitoring. Since PI changes with peripheral blood flow, it may reflect peripheral temperature gradients and, consequently, thermoregulatory responses like peripheral vasoconstriction. Studies have reported that the core-to-peripheral temperature difference correlates with peripheral PI. The findings suggest that both peripheral and core temperatures contribute to the threshold for shivering and that PI reflects the vasoconstriction induced by thermoregulatory responses that precede shivering

SUMMARY:
The goal of this observational study is to learn about the impact of intraoperative change in temperature in adult patients undergoing surgeries under general anaesthesia. The main question it aims to answer is:

Is the change in core body temperature reflected by changes in the prfusion index? Patients' core temperature, peripheral temperature and perfusion indices will be recorded throughout the span of the procedure.

DETAILED DESCRIPTION:
Perioperative hypothermia increases the risk of postoperative morbidity and mortality. Almost 50-90% of the patients experience perioperative hypothermia. This involves a decrease in core temperature to ≤ 36°C, which results in an increased rate of surgical site infection, haemorrhagic tendency, and ischemic heart disease, making it a serious perioperative complication.

Early hypothermia during general anaesthesia is mainly caused by the redistribution of body heat from the central to peripheral compartments, due to vasodilation following use of the anaesthetics. The degree of redistribution of body heat may be affected by the peripheral perfusion state, which differs across patients and results in a difference in gradient between temperature of the central and peripheral compartments. Low peripheral perfusion state can lead to low peripheral body temperature, thus lowering the overall core body temperature.

It was previously reported that the risk factors for intraoperative hypothermia are age, BMI, preoperative systolic blood pressure, heart rate, baseline core temperature, ASA-PS score, the type of anaesthesia and surgery, the duration of preparation and surgery, and ambient temperature.

Previous studies did not include the PI as a risk factor for intraoperative hypothermia. Therefore, further studies are needed to assess the relationship between PI and hypothermia to generate a more accurate predictive score of perioperative hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery under general anaesthesia
* Patients aged between 20 and 70 years old.

Exclusion Criteria:

* Patients who decline to give a written informed consent.
* Patients with psychiatric disorders that lead to inability to cooperate, speak, or read.
* BMI between <20 kg/m2 or >35 kg/m2.
* Patients undergoing emergency surgeries.
* Patients with peripheral vascular disease or rheumatoid disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery under general anesthesia in the months between April 2024 and June 2024 at Ain Shams University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
To measure the change of PI associated with change in core and peripheral body temperatures as measured by the oropharyngeal probe and the pattern of this change | Through study completion, 3 months from April 2024 to June 2024
  The PI was recorded by attaching a sensor to the patient's finger (Ultralife Pulse Oximeter JPD-500D). The baseline body temperature (T1) was measured using a Granzia GT-3 Digital thermometer. Subsequently, the PI was recorded and assessed every 15 min until completion of the surgery.

SECONDARY OUTCOMES:
To detect the change of PI with the change in temperature gradient (it is defined as the difference between the skin temperature and the core temperature) | Through study completion, 3 months from April 2024 to June 2024
To detect the incidence of a low reading of PI and the increase in serum lactate level in an arterial blood gases sample. | Through study completion, 3 months from April 2024 to June 2024
  A baseline ABG (B1) was drawn, and serum lactate value was recorded. A follow up ABG (B2) was drawn at PI values <0.2%, and serum lactate was recorded again.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No